CLINICAL TRIAL: NCT04522232
Title: Laparoscopic Hysterectomy With Prior Uterine Artery Ligation vs Conventional Laparoscopic Hysterectomy
Brief Title: Laparoscopic Hysterectomy With Prior Uterine Artery Ligation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Helwan University (Other); Cairo University (Other); Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mazen Abdel Rasheed, Principal Investigator, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uterine artery ligation in TLH
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Uterine Artery Injury; Hysterectomy
Keywords: Hysterectomy; Laparoscopy; Uterine Artery Ligation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Placebo Comparator): women that underwent conventional Total laparoscopic hysterectomy
  Interventions: Procedure: conventional Total laparoscopic hysterectomy
- group B (Experimental): women that underwent Total laparoscopic hysterectomy with prior uterine artery ligation at its origin
  Interventions: Procedure: Total laparoscopic hysterectomy with prior uterine artery ligation at its origin

INTERVENTIONS:
Procedure: conventional Total laparoscopic hysterectomy — the ascending branch of the uterine artery was identified close to the isthmus then ligated at this level, close to the uterus or coagulated, using bipolar diathermy. The utero-vesical fold was dissected and the bladder was pushed down done, thus moving the ureters laterally, which decreases the risk of including them in a suture. The vasculature of the uterus is now secured and this is evidenced by the pale color of the fundus.
  Using either bipolar diathermy or the harmonic ultracision, the cornual pedicles on one side were desiccated and cut. Also, both the uterosacral and cardinal ligaments were desiccated and cut. So that, the opposite side pedicles can be taken care of, the direction of manipulator was changed. The infundibulopelvic ligaments were desiccated and cut if it is necessary to remove both ovaries. A vaginal cuff was inserted into the vagina to identify the vault, which was then cut laparoscopically using a monopolar hook, where the specimen was completely detached.
  Arms: group A
Procedure: Total laparoscopic hysterectomy with prior uterine artery ligation at its origin — the uterine artery was dissected using the lateral approach; where dissection begins from the anterior leaf of the broad ligament. The triangle enclosed by the round ligament, external iliac artery, and infundibulopelvic ligament was opened. The areolar space was dissected and the origin of the uterine artery from the internal iliac and the ureter was identified. The uterine artery was then isolated from the surrounding structures and ligated by Hem-o-lok clips.
  then same steps as conventional Total laparoscopic hysterectomy
  Arms: group B

SUMMARY:
A randomized controlled trial was done on 127 women planned for TLH, and divided into two groups; group A includes women that underwent conventional TLH, and group B includes women that underwent TLH with prior uterine artery ligation at its origin. Both grouped were compared regarding the blood loss, operation time, intraoperative complications and post-operative follow-up.

ELIGIBILITY:
Inclusion Criteria: any benign uterine pathology such as:

* fibroid uterus
* endometrial hyperplasia with failed hormonal therapy
* DUB with failed medical and hormonal treatment
* uterine prolapse.

Exclusion Criteria:

* gynecologic malignancy
* presence of contraindications to laparoscopy.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
blood loss | during the Laparoscopy
  The total blood loss was calculated from the suction apparatus. No irrigation was used throughout the surgery until the total blood loss was calculated. Peritoneal lavage was done with normal saline solution.
operation time | during the Laparoscopy
  start time is the insertion of 10 mm telescope trocar end-time is the removal of all trocars

SECONDARY OUTCOMES:
intraoperative or postoperative complications | during the Laparoscopy and during the hospital stay (24 hours postoperative)
  intraoperative complications are that during the Laparoscopy postoperative complications are that during the hospital stay (24 hours postoperative)

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Abdel-Rasheed, Principal Investigator — National Research Centre, Egypt
Locations (1):
- Al-Azhar university hospital (new Damietta), Damietta, Egypt